CLINICAL TRIAL: NCT03200483
Title: Effects of Musical Auditory Stimulation on Autonomic Cardiac Response and Cardiorespiratory Parameters During and After Long-term Submaximal Aerobic Exercise
Brief Title: Musical Auditory Stimulation and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, PHD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2200/11
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Autonomic Nervous System; Cardiorespiratory Parameters
Keywords: Autonomic Nervous System; Aerobic exercise; Recuperation; Music

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Control Protocol (Experimental): The volunteer will perform the exercise and recovery exposed to silence
  Interventions: Other: Control Protocol
- Classical Music Protocol (Experimental): The volunteer will perform the exercise and recovery exposed to classical music
  Interventions: Other: Classical Music Protocol
- Rock Music Protocol (Experimental): The volunteer will perform the exercise and recovery exposed to rock musical style
  Interventions: Other: Rock Music Protocol

INTERVENTIONS:
Other: Control Protocol — In this period the volunteers were at rest, in the supine position for 15 minutes, followed by 30 minutes of aerobic exercise on a treadmill (five minutes at a speed of 6.0 km / h followed by 25 minutes with 60% of Vmax + 1% grade) and then a recovery period lasting 60 minutes (three minutes standing on the treadmill followed by 57 minutes in the supine position). The volunteers were instructed to remain awake during all the protocol and this was verified and monitored by one of the researchers.
  Arms: Control Protocol
Other: Classical Music Protocol — Volunteers accomplished the same activities of the control protocol, but with exposure to classical music during exercise and recovery.
  Arms: Classical Music Protocol
Other: Rock Music Protocol — Volunteers accomplished the same activities of the control protocol, but with exposure to rocky musical style during exercise and recovery.
  Arms: Rock Music Protocol

SUMMARY:
Check the effects of musical auditory stimulation on the autonomic modulation and cardiorespiratory parameters during and after aerobic exercise. Hypothesized that classical music can increase recovery velocity after exercise and rock style music can generate a delay in the recovery velocity of the cardiorespiratory parameters and in the cardiac autonomic response.

DETAILED DESCRIPTION:
To implement the experimental protocol, all volunteers were informed to not ingest alcoholic or caffeine-based drinks for 12 hours before the experimental procedure; consuming light meal only two hours before and avoid any vigorous physical exertion 24 hours before the testing.

The experimental procedures were divided into three segments, all performed on a treadmill, with a minimum interval of 48 hours between them in order to allow the volunteers to recover. The protocols running time was always set between 5:30 PM and 9:30 PM, to avoid circadian influences. In addition to these, temperature was fixed between 23 ° C and 24 ° C and humidity between 60% and 70%.

Before the first phase of the experimental protocol the volunteers were approved and the investigators obtained body mass by means of a digital scale (Plenna, TIN 00139 Maxima, Brazil) then height, by means of a stadiometer (ES 2020 - Sanny, Brazil). The comparable stages of the experimental protocol were undertaken:

I) Maximal exercise test: the investigators undertook this to record the maximum velocity (Vmax) reached by the volunteer. This was then applied to indirectly determine the anaerobic threshold via the Conconi threshold. Intensity of 60% of the Vmax obtained in the test was lesser than that found in the anaerobic threshold, and this intensity was enforced to perform subsequent steps;

II) Control Protocol (CP): In this period the volunteers were at rest, in the supine position for 15 minutes, followed by 30 minutes of aerobic exercise on a treadmill (five minutes at a speed of 6.0 km / h followed by 25 minutes with 60% of Vmax + 1% grade) and then a recovery period lasting 60 minutes (three minutes standing on the treadmill followed by 57 minutes in the supine position). The volunteers were instructed to remain awake during all the protocol and this was verified and monitored by one of the researchers.

III) Music Protocol (MP): Volunteers accomplished the same activities of the CP, but with exposure to musical auditory stimulation during exercise and recovery.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* Smokers, alcoholics, subjects with cardiovascular, respiratory and neurological disorders known or other pathological conditions that prevented the achievement of protocols will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Music effects on heart rate variability based on time domain | 90 minutes
Music effects on heart rate variability based on frequency domain | 90 minutes
Music effects on heart rate variability based on Chaos domain | 90 minutes
Blood pressure (mmHg) | 90 minutes
Heart rate (beats per minute) | 90 minutes
Respiratory rate (per minute) | 90 minutes
Oxygen saturation pulse (SpO2) | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos Marques Vanderlei, ph.D, Principal Investigator — Universidade Estadual Paulista - UNESP